CLINICAL TRIAL: NCT00933608
Title: Effects of Memantine on the Magnetic Resonance Spectroscopy (MRS) Measures of Neuronal Integrity in Subjects at Risk for Alzheimer's Disease
Brief Title: Effects of Memantine on Magnetic Resonance (MR) Spectroscopy in Subjects at Risk for Alzheimer's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Lidia Glodzik, Assistant Research Professor, NYU Langone Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NAM-MD-68
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Results first posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Alzheimer's Disease
Keywords: subjective memory complaints; cognitively healthy; family history; AD
MeSH Terms: conditions — Alzheimer Disease | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- memantine (Experimental): after a period of gradual dose increase from 5 mg/day, participants will be asked to take memantine (20mg/day) for 16 weeks 10 mg in the morning, 10 mg at night
  Interventions: Drug: memantine
- Placebo (Placebo Comparator): dose increase to match active drug, after that 1 tablet in the morning, 1 tablet at night, to match active drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: memantine — participants will be asked to take memantine (20mg/day) for 16 weeks
  Other Names: Namenda
  Arms: memantine
Drug: Placebo — participants will be asked to take 2 tablets per day to match active drug
  Arms: Placebo

SUMMARY:
Recent data show that marked cell damage precedes the clinical manifestation of Alzheimer's disease (AD). Hence, targeting populations at risk with pharmacological interventions is a possible strategy to lessen the burden of the disease. Cognitively normal individuals with subjective memory complaints (SMC) manifest biological characteristics consistent with early AD and are at risk for future cognitive decline. Family history of AD also constitutes a risk. In a previous study the investigators showed that memantine slows down the accumulation of phosphorylated tau in normal SMC subjects. Using a multivoxel high field MR spectroscopy (MRS) technique, the investigators also demonstrated that memantine decreased hippocampal glutamate. Both these findings may be consistent with the drug's anti-excitotoxic activity. In this new project the investigators propose to treat a sample of 12 presymptomatic individuals at risk (SMC and family history of AD) with memantine. This will be a double blind, placebo controlled study with a control group (12 non-treated subjects). The investigators will determine whether the effects of memantine as assessed by cognitive performance and MRS are present after 4 months of treatment and persist 2 months after discontinuation. MRS will be used to evaluate the effect of memantine on levels of the neurotransmitter glutamate and neuronal viability marker N-acetylaspartate (NAA) in the hippocampus. The investigators will test the following hypotheses:

1. In subjects with SMC, memantine has modifying effects on brain biochemistry as reflected in MRS reductions in glutamate (reduced excitotoxicity) and increases in NAA (neuronal integrity).
2. The effects of the drug persist (as a marker of sustained neuroprotection) and can be measured 2 months after discontinuation of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* presence of subjective memory complaints without objective evidence of impaired cognition
* family history of Alzheimer's disease

Exclusion Criteria:

* major depression
* Parkinson's disease
* stroke
* seizures
* uncontrolled diabetes or hypertension
* current benzodiazepine use
* substance abuse
* contraindication for MRI
* contraindications for memantine

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lidia Glodzik, MD PhD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU School of Medicine, Dept. of Psychiatry, Center for Brain Health, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study was carried out at the NYU Center for Brain Health and Aging and Dementia Center, between May 2010 and October 2011.
Groups:
- Memantine: memantine : participants will be asked to take memantine (20mg/day) for 16 weeks
- Placebo: participants were taking 1 tablet twice a day to match memantine arm
Period: Overall Study
Arm/Group | Memantine | Placebo
Started | 7 | 10
Completed | 2 | 8
Not Completed | 5 | 2
Not completed — Adverse Event | 4 | 2
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Memantine | Placebo | Total
Number analyzed (Participants) | 7 | 10 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 5
  >=65 years | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (5.7) | 69.7 (8.2) | 69.7 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 1 | 5 | 6
Region of Enrollment [Number; unit: participants]
  United States | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: N-acetylaspartate
Description: The change in N-acetylaspartate (NAA) measured with magnetic resonance spectroscopy (MRS) is the primary outcome measure. NAA is a metabolite found predominately in neuronal cells, and its amount indicates tissue well being (the higher the better). In MRS studies NAA (and other metabolites like choline or myoinositol) are presented as a ratio to creatine (Cr) also measured by MRS. The concentration of creatine does not change is used as an internal standard. The ratio NAA/Cr is unitless. In summary, the measurable outcome will be the NAA/Cr ratio change from pre-to post treatment.
Time Frame: baseline (pre-treatment) and 4 months (post-treatment)
Population: This is an intention to treat analysis, based on initial treatment assignment.
Measure: Mean (Standard Deviation); unit: NAA/creatine Ratio
Groups:
- Placebo: participant will be taking 1 tablet twice a day to match active arm
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 4 | 9
NAA/creatine Ratio
  pre-treatment | 1.35 (.38) | 1.86 (.43)
  post-treatment | 1.58 (.005) | 1.26 (.49)

ADVERSE EVENTS:
Arm/Group | Memantine | Placebo
Serious Adverse Events (participants affected / at risk) | 1/7 | 1/10
Other Adverse Events (participants affected / at risk) | 3/7 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Memantine (N=7) | Placebo (N=10)
loss of consciousness (General disorders) | 1 | 0
severe anemia (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Memantine (N=7) | Placebo (N=10)
skin rash (Skin and subcutaneous tissue disorders) | 1 | 0
dizziness (Ear and labyrinth disorders) | 1 | 0
high blood presure (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No